CLINICAL TRIAL: NCT03053700
Title: Intense Pulsed Light as an Adjunctive to Bromonidine for the Treatment of Rosacea- a Prospective Study
Brief Title: Intense Pulsed Light as an Adjunctive to Bromonidine for the Treatment of Rosacea
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: During study new treatments were available, which may be more effective than proposed study treatment.
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0682-16RMC
Record Dates: First submitted 2017-02-06; First posted 2017-02-15 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2018-09

CONDITIONS: Rosacea
Keywords: Rosacea, Bromonidine, intensed pulse light
MeSH Terms: conditions — Rosacea | interventions — Gels

STUDY DESIGN:
Intervention Model Description: This is an interventional, prospective single blinded study. Patients would be treated with full face application of bromonide 0.33% gel once daily for three months. In addition half of the patients' face would be subjected to three IPL treatment sessions three weeks apart from each other.
Who Masked: Outcomes Assessor
Masking Description: Physicians will perform assessment of clinical outcome, using clinical photographs .These physicians will be blinded to which half of the face was treated with intense pulsed light.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with bromonide 0.33% gel (Active Comparator): Patients would be treated with full face application of bromonide 0.33% gel once daily for three months. Half of the patients' face would recieve this treatment alone.
  Interventions: Drug: Bromonide 0.33% gel
- Treatment with bromonide 0.33% gel & IPL (Active Comparator): Patients would be treated with full face application of bromonide 0.33% gel once daily for three months. Half of the patients' face would be subjected to three IPL treatment sessions three weeks apart from each other.
  Interventions: Drug: Bromonide 0.33% gel; Device: Intense Pulsed Light (M22)

INTERVENTIONS:
Drug: Bromonide 0.33% gel — Patients would be treated with full face application of bromonide 0.33% gel once daily for three months.
Device: Intense Pulsed Light (M22) — Half of the patients' face would be subjected to three IPL treatment sessions three weeks apart from each other.
  Arms: Treatment with bromonide 0.33% gel & IPL

SUMMARY:
This is an interventional and prospective study. The study is designed to evaluate the additional benefits of a combination of IPL treatment and local application of Bromonide 0.33% gel in the treatment of erythematotelangiectatic (ETR) and papulopustular (PPR).

DETAILED DESCRIPTION:
Patients would be treated with full face application of bromonide 0.33% gel once daily for three months. In addition half of the patients' face would be subjected to three IPL treatment sessions three weeks apart from each other.

ELIGIBILITY:
Inclusion Criteria:

* patient (male or female) must be over 18 yaers old of age and fulfil one of the following:

  1. Suffer from ETR
  2. Suffer from PPR
  3. Suffer from a combination of ETR and PPR.

Exclusion Criteria:

* 1.Under 18 years old of age. 2.Pregnant women. 3.Systemic treatment of rosacea at the previous six months before enrollment. 4.Topical treatment of rosacea at the previous one month before enrollment. 5.Phymatous or occular rosacae.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
patient self-assessment questionaires score change | three months after initiation of treatment compared to Baseline
  Patient will assess disease change on 5 points scale (0=no improvement, 1=0-25% improvement, 2=26-49% improvement, 3=50-74% improvement, 4= 75-100% improvement.
Physicians' unblinded score assessment | three months after initiation of treatment compared to Baseline
  Physician will assess disease change on 5 points scale (0=no improvement, 1=0-25% improvement, 2=26-49% improvement, 3=50-74% improvement, 4= 75-100% improvement.
Physicians' unblinded score assessment | six months after initiation of treatment compared to Baseline
  Physician will assess disease change on 5 points scale (0=no improvement, 1=0-25% improvement, 2=26-49% improvement, 3=50-74% improvement, 4= 75-100% improvement.
patient self-assessment questionaires score change | six months after initiation of treatment compared to Baseline
  Patient will assess disease change on 5 points scale (0=no improvement, 1=0-25% improvement, 2=26-49% improvement, 3=50-74% improvement, 4= 75-100% improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Assi Levi, Dr., Principal Investigator — Rabin Medical center, Petach Tikva
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No